CLINICAL TRIAL: NCT03718897
Title: Identification of Prognostic Gene Mutations in Biliary Tract Cancer Using Whole Genome Sequencing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ji Kon Ryu (Other)
Responsible Party: Sponsor-Investigator, Ji Kon Ryu, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: 1808-056-964
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Whole genome sequencing of biopsy specimen of biliary tract cancer
  2. Peripheral blood circulating tumor DNA in patients with biliary tract cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic retrograde cholangiopancreatogram — Biopsy specimens are attained via endoscopic retrograde cholangiopancreatogram in patients with suspicious biliary tract cancer.

SUMMARY:
The purpose of this study is to investigate genetic mutations affecting prognosis using whole genome sequencing in patients with biliary tract cancer.

DETAILED DESCRIPTION:
Recently, as genome technology such as next-generation sequencing has progressed, precision medicine using genetic analysis in lung cancer, colorectal cancer, and melanoma has been actively studied. The need for such precision medicine is also increasing in biliary tract cancer patients. Although whole genome sequencing is relatively costly, it is known to provide more accurate information than other methods such as exome analysis and RNA sequencing in identifying promoter mutations, regulatory regions, and structural variants. Pancreatic cancer and melanoma have been studied by whole genome sequencing, but there is no previous study using whole genome sequencing method in biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with biliary tract cancer via endoscopic retrograde cholangiopancreatogram

Exclusion Criteria:

* Pregnancy
* Other active tumors within 5 years
* Coagulopathy
* Severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the study period, all patients who were diagnosed with biliary tract cancer via endoscopic retrograde cholangiopancreatogram at Seoul National University Hospital will be enrolled. The investigators will perform whole genome sequencing of biopsy specimens from patients with biliary tract cancer and analyze the gene mutations associated with patient survival. And additionally, the presence or absence of blood circulating tumor DNA and associated gene mutation will be analyzed.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-09-02 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 48 months
  Comparisons of overall survival rates between patients with gene mutations and without.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Kon Ryu, MD, phD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No